CLINICAL TRIAL: NCT05782959
Title: An Open-Label, Dose-Escalation, Non-comparative Clinical Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of BCD-245 (JSC BIOCAD, Russia) Administered Intravenously to Subjects With Neuroblastoma
Brief Title: Phase 1 Study of BCD-245 in Subjects With Neuroblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BCD-245-1
Record Dates: First submitted 2023-02-16; First posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-02

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): BCD-245 (anti-GD-2 monoclonal antibody), dose 1
  Interventions: Biological: BCD-245
- Cohort 2 (Experimental): BCD-245 (anti-GD-2 monoclonal antibody), dose 2
  Interventions: Biological: BCD-245
- Cohort 3 (Experimental): BCD-245 (anti-GD-2 monoclonal antibody), dose 3
  Interventions: Biological: BCD-245
- Cohort 4 (Experimental): BCD-245 (anti-GD-2 monoclonal antibody), dose 4
  Interventions: Biological: BCD-245

INTERVENTIONS:
Biological: BCD-245 — BCD-245 is administered as prolonged intravenous infusions during each cycle

SUMMARY:
The aim of the study is to investigate the safety, pharmacokinetics, pharmacodynamics, and immunogenicity of BCD-245 after its single and multiple intravenous infusions at escalating doses in subjects with relapsed/refractory neuroblastoma.

DETAILED DESCRIPTION:
The study includes 2 stages: 1) Data collection and safety analysis for the first four subjects 12 years of age and older from Cohort 1 2) Data collection and analysis of safety, pharmacokinetics, pharmacodynamics and immunogenicity in all cohorts (Cohorts 1-4).

The design of this Phase I study is based on standard 3 + 3 design approaches. Cohort 1 includes 4 subjects aged 12 years old and older, and 2 subjects aged 3 years old and older. Cohorts 2-4 include 3-6 subjects aged 3 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 years and older (12 years and older for the first four subjects) at the time of signing the informed consent form
* Established diagnosis of neuroblastoma (confirmed by the study site laboratory where the subject will be treated) based on: a) histological examination of the tumor tissue (with or without immunohistochemistry) or b) presence of typical tumor agglomerates in the bone marrow and/or meta-iodobenzylguanidine-accumulating focus (foci) and an increase in the level of catecholamine metabolites in serum and/or urine
* Relapsed or refractory neuroblastoma resistant to the anti-relapse therapy adopted at the study site
* Satisfactory performance status (>70 on the Lansky or Karnofsky scale)
* Life expectancy >8 weeks

Exclusion Criteria:

* Indications for radiation therapy, surgical intervention for the primary disease at screening
* Isolated CNS relapse of neuroblastoma
* Planned use of any anticancer drugs concomitantly with BCD-245 in this clinical trial
* The need for continuous use of anticonvulsants
* Clinically significant neurological deficit or grade >2 peripheral neuropathy (CTCAE 5.0)
* The need or probable need for systemic continuous use of glucocorticosteroids or other immunosuppressive drugs
* Signs of respiratory distress (dyspnea at rest and oxygen saturation <94% without oxygen supplementation)
* Any severe organ dysfunction (> CTCAE 5.0 severity grade 2) at screening, except for hematological abnormalities.
* Body weight less than 10 kg.
* Subject receiving anti-GD2 monoclonal antibody therapy within 6 weeks or less prior to intended study drug infusion

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with adverse reactions | 52 weeks
Proportion of subjects with serious adverse reactions | 52 weeks
Proportion of subjects with adverse reactions of grade 3 or higher according to CTCAE 5.0 | 52 weeks
Proportion of therapy discontinuations due to adverse reactions | up to 4 weeks

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from time zero to t (AUC 0-t) | up to 4 weeks
Area under the plasma concentration versus time curve from zero to time infinity (AUC 0-∞) | up to 4 weeks
Peak plasma concentration (Cmax) | up to 4 weeks
Time of peak plasma concentration (Tmax) | up to 4 weeks
Half-life (T1/2) | up to 4 weeks
  Half-life is the time taken to decrease the plasma concentration of a drug to one-half its original value
Volume of distribution (Vd) | up to 4 weeks
Mean steady-state peak plasma concentration (Cmax) | 20 weeks
Pre-dose trough concentration (Ctrough) | 20 weeks
Counts of lymphocytes and CD56+CD16+ (cytokine-secreting and cytotoxic) NK cells | 52 weeks
Whole blood cytolytic activity test | 52 weeks
Proportion of subjects with anti-BCD-245 BAbs and NAbs | 52 weeks

OTHER OUTCOMES:
Overall response rate | 52 weeks
  Includes complete response, very good partial response, partial response
Duration of response | 52 weeks
Time to response | 52 weeks
Event-free survival | 52 weeks
Overall survival | 52 weeks

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Dmitry Rogachev National Medical Research Center Of Pediatric Hematology, Oncology and Immunology, Moscow
  - Russian Cancer Research Center named after N.N. Blokhin "of the Ministry of Health of the Russian Federation, Moscow
  - Raisa Gorbacheva Memorial Research Institute of Children Oncology, Hematology and Transplantation, Saint Petersburg